CLINICAL TRIAL: NCT05043779
Title: Is Preoperative Awake Airway Nasoendoscopy A Good Tool To Predict The Expected Difficult Airway In Obese Patients?
Brief Title: Evaluation of Preoperative Nasoendoscopy to Predict Difficult Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRC-01-19-107
Record Dates: First submitted 2021-07-28; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-07

CONDITIONS: Difficult or Failed Intubation; Obesity, Morbid
Keywords: Nasoendoscopy,; Obesity,; Difficult intubation
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Awake Airway Nasoendoscopy (Other): only one arm
  Interventions: Procedure: Awake Airway Nasoendoscopy

INTERVENTIONS:
Procedure: Awake Airway Nasoendoscopy — Preoperative Awake Airway Nasoendoscopy of upper airway

SUMMARY:
Despite the availability of different methods for airway assessment, unexpectedly difficult intubations occur at a frequency of up to 15%. A variety of pre-intubation clinical screening tests have been advocated to predict difficult laryngoscopy and airway but their usefulness is limited in obese patients.

Could awake invasive airway assessment be more predictive for difficult airways in obese patients? The use of nasendoscopy assessment for the airway could be a useful additional invasive tool to predict the difficult airway in obese

DETAILED DESCRIPTION:
Predictors of difficult laryngoscopy and intubation may be less useful or irrelevant when there is a plan for video laryngoscopes (VL) intraoperative. VL improves laryngeal view in most patients, Their use achieves a high success rate for intubation of patients with predicted difficult intubation, and those who have failed direct laryngoscopy[6]. In a study of over 2000 (VL) video laryngoscopies intubations, Mallampati's score did not correlate with failed intubation. The strongest predictor of failure was neck pathology, including the presence of a surgical scar, radiation changes, or mass. In another study, risk factors for difficult VL intubation after direct laryngoscopy were Cormack-Lehane grade 3 or 4 views with direct laryngoscopy, short sternothyroid distance, and high upper lip bite test score. Obesity is a recognized risk factor for difficulty with airway management. An audit of major complications of airway management (NAP4) from over three million anesthetics in the United Kingdom found twice as many case reports of major complications in obese patients, especially in the morbidly obese.

It is less clear whether obesity increases the risk of difficult laryngoscopy or intubation. Some studies suggest that obesity is a risk factor for both difficult mask ventilation and difficult laryngoscopy, while other studies suggest that with proper positioning and preparation, ventilation and laryngoscopy are not difficult [12,13]. Wilson's score is an important development in predictivity of airway difficulties, Wilson's in his study (1988) attempted to deductively identify patients for whom intubation will be difficult.

This study aims to demonstrate the use of preoperative awake fibreoptic examination

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-60 years of age either male or female with (ASA I, II or III ), scheduled for a bariatric procedure with a body mass index (BMI) greater than 35 K/M2, will be enrolled

Exclusion Criteria:

* Patients on the tracheostomy tube
* Patients who are unable to give consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Naso-endoscopy views from nose to larynx in obese patients using NOHL score during pre-operative assessment. | During pre-operative assessment.
  Findings will be recorded and scored according to NOHL (N=nose, O= oral, H= hypopharynx and L= Larynx ) every parameter takes a score from 1- 4 during pre-operative assessment.(the maximum values score = 16 and the minimum = 4)

SECONDARY OUTCOMES:
Measurement of neck circumference in Centimeter | During pre-operative assessment.
  This will be measured by centimeter during pre-operative assessment using a ruler
Mouth opening measurement by Centimeter | During pre-operative assessment.
  This will be measured by centimeter between incisors during pre-operative assessment using a ruler and documented by Centimeter
Thyro-mental distance measurement by Centimeter | During pre-operative assessment.
  This will be measured by centimeter from thyroid cartilage to patient's chin during pre-operative assessment using a rule
Difficult mask ventilation score (1 -3) | During Induction of anesthesia
  Degree of Difficulty in mask ventilation will be graded (1= easy, 2= difficult or 3=impossible) during induction of general anaesthesia
Cormak-Lehans grade during induction of anaesthesia | During intubation
  Cormak-Lehans Score will graded during endotracheal intubation and exposure of the larynx. (Grade 1= easy intubation while grade Grade 4= very difficult intubation)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Shallik, M.D., Principal Investigator — Hamad Medical Corporation - HMC
Locations (1):
- ACC, Hamad Medical Corporation, Doha, Doah, Qatar

IPD SHARING:
Plan to Share IPD: Yes
We will share after IRB approval
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After approval IRB directly
Access Criteria: Through Website

REFERENCES:
- [Result] Butler PJ, Dhara SS. Prediction of difficult laryngoscopy: an assessment of the thyromental distance and Mallampati predictive tests. Anaesth Intensive Care. 1992 May;20(2):139-42. doi: 10.1177/0310057X9202000202. PMID 1595845
- [Result] Janssens M, Hartstein G. Management of difficult intubation. Eur J Anaesthesiol. 2001 Jan;18(1):3-12. doi: 10.1046/j.0265-0215.2000.00777.x. PMID 11270007
- [Result] Qudaisat IY, Al-Ghanem SM. Short thyromental distance is a surrogate for inadequate head extension, rather than small submandibular space, when indicating possible difficult direct laryngoscopy. Eur J Anaesthesiol. 2011 Aug;28(8):600-6. doi: 10.1097/EJA.0b013e328347cdd9. PMID 21610502
- [Result] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Result] Tremblay MH, Williams S, Robitaille A, Drolet P. Poor visualization during direct laryngoscopy and high upper lip bite test score are predictors of difficult intubation with the GlideScope videolaryngoscope. Anesth Analg. 2008 May;106(5):1495-500, table of contents. doi: 10.1213/ane.0b013e318168b38f. PMID 18420866
- [Result] Samsoon GL, Young JR. Difficult tracheal intubation: a retrospective study. Anaesthesia. 1987 May;42(5):487-90. doi: 10.1111/j.1365-2044.1987.tb04039.x. PMID 3592174
- [Result] Sun DA, Warriner CB, Parsons DG, Klein R, Umedaly HS, Moult M. The GlideScope Video Laryngoscope: randomized clinical trial in 200 patients. Br J Anaesth. 2005 Mar;94(3):381-4. doi: 10.1093/bja/aei041. Epub 2004 Nov 26. PMID 15567809
- [Result] Lundstrom LH, Moller AM, Rosenstock C, Astrup G, Wetterslev J. High body mass index is a weak predictor for difficult and failed tracheal intubation: a cohort study of 91,332 consecutive patients scheduled for direct laryngoscopy registered in the Danish Anesthesia Database. Anesthesiology. 2009 Feb;110(2):266-74. doi: 10.1097/ALN.0b013e318194cac8. PMID 19194154
- [Result] Heinrich S, Birkholz T, Ihmsen H, Irouschek A, Ackermann A, Schmidt J. Incidence and predictors of difficult laryngoscopy in 11,219 pediatric anesthesia procedures. Paediatr Anaesth. 2012 Aug;22(8):729-36. doi: 10.1111/j.1460-9592.2012.03813.x. Epub 2012 Feb 20. PMID 22340664
- [Result] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Result] Brodsky JB, Lemmens HJ, Brock-Utne JG, Vierra M, Saidman LJ. Morbid obesity and tracheal intubation. Anesth Analg. 2002 Mar;94(3):732-6; table of contents. doi: 10.1097/00000539-200203000-00047. PMID 11867407
- [Result] Wilson ME, Spiegelhalter D, Robertson JA, Lesser P. Predicting difficult intubation. Br J Anaesth. 1988 Aug;61(2):211-6. doi: 10.1093/bja/61.2.211. PMID 3415893
- [Result] Vicini C, De Vito A, Benazzo M, Frassineti S, Campanini A, Frasconi P, Mira E. The nose oropharynx hypopharynx and larynx (NOHL) classification: a new system of diagnostic standardized examination for OSAHS patients. Eur Arch Otorhinolaryngol. 2012 Apr;269(4):1297-300. doi: 10.1007/s00405-012-1965-z. Epub 2012 Feb 19. PMID 22350494
- [Result] Soares MC, Sallum AC, Goncalves MT, Haddad FL, Gregorio LC. Use of Muller's maneuver in the evaluation of patients with sleep apnea--literature review. Braz J Otorhinolaryngol. 2009 May-Jun;75(3):463-6. doi: 10.1016/S1808-8694(15)30667-4. PMID 19649500